CLINICAL TRIAL: NCT06177964
Title: Randomized Phase 2 Clinical Trial of Repeated Intratumoral and Cervical Perilymphatic Lerapolturev Injections Versus Lomustine in Recurrent Glioblastoma (GBM)
Brief Title: Lerapolturev (PVSRIPO) in GBM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Darell Bigner (Other)
Collaborators: Istari Oncology, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Darell Bigner, Professor of Neurosurgery, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00113584
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Supratentorial Glioblastoma
Keywords: Lerapolturev; PVSRIPO; Lomustine; Shoaf; Glioblastoma; Glioma; Pro00113584; Duke; Istari Oncology; Intratumoral injection; Cervical Perilymphatic injection
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lerapolturev Arm (Stage 1) (Experimental): Lerapolturev (intratumoral) will be dosed by Convection Enhanced Delivery (CED), infused twice, 4 days apart, in the remaining disease of recurrent Glioblastoma (rGBM) subjects following maximal safe resection of the disease recurrence.
  To assess treatment response and/or immunologic responses in the brain, a tissue biopsy of the area infused will be recommended 5 weeks (± 1 week) after the 2nd lerapolturev infusion via CED, in the event that changes suggestive of tumor progression are seen on the MRI obtained 4-5 weeks after the 2nd lerapolturev infusion via CED.
  .
  Interventions: Drug: Lerapolturev
- Lerapolturev Arm (Stage 2 - Arm 1) (Experimental): Lerapolturev (intratumoral) will be given by Convection Enhanced Delivery (CED), infused twice, 4 days apart, in the remaining disease of recurrent Glioblastoma (rGBM) subjects following maximal safe resection of their disease recurrence. This will be followed by subcutaneous injections of lerapolturev in the cervical perilymphatic (CPL) area on the same side as their tumor, weekly for 4 weeks and afterward every 3 weeks for about a year.
  Interventions: Drug: Lerapolturev
- Lomustone (Stage 2 Arm 2) (Active Comparator): Following maximal safe resection of their tumor recurrence subjects will receive Lomustine as a single oral dose of 110 mg/m2 every six weeks for up to 9 cycles.
  Interventions: Drug: Lomustine Pill

INTERVENTIONS:
Drug: Lerapolturev — Lerapolturev (intratumoral) will be dosed at 2x108 TCID50 in 3.0 mL x 2 doses (total dose 4x108 TCID50) by Convection Enhanced Delivery.
  For the patients randomized to the lerapolturev Arm 1 of Stage 2, seven days (±2 days) following completion of the 2nd intratumoral infusion of lerapolturev, patients will begin cervical perilymphatic subcutaneous injection of lerapolturev at a dose of 2 x 108 TCID50 (in 0.5 ml diluent) around the cervical lymph node chain ipsilateral to the intracranial tumor.
  Arms: Lerapolturev Arm (Stage 1); Lerapolturev Arm (Stage 2 - Arm 1)
Drug: Lomustine Pill — Lomustine will be given as a single oral dose of 110 mg/m2 every six weeks for up to 9 cycles.
  Arms: Lomustone (Stage 2 Arm 2)

SUMMARY:
The purpose of this research study is to determine the safety and efficacy of administering two doses of lerapolturev in residual disease (within tumor margins) after surgery, followed later by repeated injections of lerapolturev in the subcutaneous area (under the skin) around the lymph nodes of the head and neck for adult patients diagnosed with recurrent glioblastoma at the Preston Robert Tisch Brain Tumor Center (PRTBTC) at Duke.

DETAILED DESCRIPTION:
The study will be conducted in two stages: Approximately twelve patients with recurrent supratentorial glioblastoma will enroll in stage 1.

Stage 1 is a safety lead-in which will assess the safety of lerapolturev when infused twice, 4 days apart, via Convection Enhanced Delivery (CED) in the residual disease of recurrent Glioblastoma (GBM) patients following maximal safe resection of the enhancing/necrotic portion of the disease recurrence.

A tissue biopsy of the area infused will be recommended 5 weeks (± 1 week) after the 2nd lerapolturev infusion via CED, if imaging changes suggest tumor progression vs. immune effect on the MRI obtained 4-5 weeks after the 2nd lerapolturev infusion via CED.

Stage 2 is a Phase 2 randomized clinical trial to compare the efficacy and safety of two treatment regimens for recurrent GBM patients who undergo maximal safe resection for their recurrence. Approximately eighty patients with recurrent supratentorial glioblastoma will enroll in stage 2 of the study.

Stage 2 has 2 arms and is randomized, like the flip of a coin. Arm 1 is Lerapolturev and Arm 2 is Lomustine. After the recurrent tumor has been removed by surgery, subjects will be randomly assigned to receive either the FDA-approved chemotherapy (lomustine) or the study drug (lerapolturev). Subjects receive lerapolturev infused in the residual disease via CED twice, 4-day apart. About 1 week after the 2nd lerapolturev infusion, subjects will start subcutaneous (under the skin) injections of lerapolturev into the area of the cervical lymph nodes (head and neck) nearest to their tumor weekly for 4 weeks and afterward every 3 weeks for about a year.

Subjects assigned to receive lomustine will begin taking it 3-4 weeks after surgery to remove their recurrent tumor. One prescribed dose of lomustine will be taken no more than once every 6 weeks, for no more than 1 year or up to 9 cycles.

Subjects will be followed for serious adverse events (side effects) for 30 days after stopping the study. Subjects' medical records will be reviewed for the remainder of their life, in order to collect data on subsequent treatments, disease progression, tumor size/volume, and survival.

There are risks to the study drug, lerapolturev, and the chemotherapy drug, lomustine. The most common risks of lerapolturev are headache, seizure, weakness on one side of the body, difficulty thinking or processing, difficulty receiving or responding to sensory information, fatigue, and difficulty speaking or comprehending. Risks associated with infusion procedure include mild discomfort at the infusion site, bleeding in the brain, pain, infection, and swelling of the brain. The study drug and procedures used together could also potentially cause more serious side effects. The most common risks of lomustine are changes in your red blood cell count, changes in platelets, changes in your liver, feeling confused and tired, poor appetite, and loss of ability to conceive or father a child.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old at the time of entry into the study.
2. Histopathologically confirmed recurrent supratentorial glioblastoma (WHO grade 4) (high grade glioma with molecular features of glioblastoma will be eligible).
3. Karnofsky Performance Score (KPS) ≥ 70%
4. Hemoglobin ≥ 9 g/dl prior to biopsy
5. Platelet count ≥ 100,000/µl unsupported is necessary for eligibility on the study; however, because of risks of intracranial hemorrhage with catheter placement, platelet count ≥ 125,000/µl is required for the patient to undergo biopsy and catheter insertion, which can be attained with the help of platelet transfusion.
6. Neutrophil count ≥ 1000 prior to biopsy
7. Creatinine ≤ 1.5 x normal range prior to biopsy
8. Total bilirubin ≤ 1.5 x ULN prior to biopsy (Exception: Participant has known or suspected Gilbert's Syndrome for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable.)
9. AST/ALT ≤ 2.5 x ULN
10. Prothrombin and Partial Thromboplastin Times ≤ 1.2 x normal prior to biopsy. Patients with prior history of thrombosis/embolism are allowed to be on anticoagulation, understanding that anticoagulation will be held in the perioperative period per the neurosurgical team's recommendations. Low molecular weight heparin (LMWH) is preferred. If a patient is on warfarin, the international normalized ratio (INR) is to be obtained and value should be below 2.0 prior to biopsy.
11. At the time of biopsy, prior to administration of the 1st infusion of lerapolturev via CED, the presence of recurrent tumor must be confirmed by histopathological analysis.
12. Able to undergo brain MRI with and without contrast
13. Prior CDC-recommended vaccination series against PV and has received a boost immunization with trivalent Poliovirus Vaccine Inactivated (IPOL®) (Sanofi-Pasteur SA) at least 1 week, but less than 6 weeks, prior to administration of lerapolturev. Note: Patients who are unsure of their prior vaccination status must provide evidence of anti-PV immunity prior to enrollment, as applicable.
14. Patient or partner(s) meets one of the following criteria:

    1. Non-childbearing potential (i.e., not sexually active, physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile, or any male who has had a vasectomy). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Postmenopausal for purposes of this study is defined as 1 year without menses.; or
    2. Childbearing potential and agrees to use one of the following methods of birth control: approved hormonal contraceptives (e.g. birth control pills, patches, implants, or infusions), an intrauterine device, or a barrier method of contraception (e.g., a condom or diaphragm) used with spermicide.
15. A signed informed consent form approved by the Institutional Review Board (IRB) will be required for patient enrollment into the study. Patients must be able to read and understand the informed consent document and must sign the informed consent indicating that they are aware of the investigational nature of this study

Exclusion Criteria:

1. Females who are pregnant or breast-feeding
2. Patients with an impending, life-threatening cerebral herniation syndrome, based on the assessment of the study neurosurgeons or their designate
3. Patients with severe, active co-morbidity, defined as follow:

   1. Patients with an active infection requiring intravenous treatment or having an unexplained febrile illness (Tmax > 99.5°F/37.5°C)
   2. Patients with known immunosuppressive disease or known human immunodeficiency virus infection
   3. Patients with unstable or severe intercurrent medical conditions such as severe heart disease (New York Heart Association Class 3 or 4)
   4. Patients with known lung (forced expiratory volume in the first second of expiration (FEV1) < 50%) disease or uncontrolled diabetes mellitus
4. Known albumin allergy
5. History of agammaglobulinemia
6. Patients may not have received chemotherapy or bevacizumab ≤ 4 weeks [except for nitrosourea (6 weeks), or metronomic dosed chemotherapy such as daily etoposide or cyclophosphamide (1 week)] prior to starting the study drug unless patients have recovered from side effects of such therapy
7. Patients may not have received immunotherapy ≤ 4 weeks prior to starting the study drug unless patients have recovered from side effects of such therapy
8. Patients may not have received treatment with tumor treating fields (e.g., Optune®) ≤ 1 week prior to starting the study drug
9. Patients may not be less than 12 weeks from radiation therapy, unless progressive disease outside of the radiation field or 2 progressive scans at least 4 weeks apart or histopathologic confirmation
10. Patients who have not completed all standard of care treatments, including surgical procedure and radiation therapy (Please note: For patients under 65 years old, standard radiation therapy is typically at least 59 Gy in 30 fractions over 6 weeks. For patients 65 years or older, standard RT is often reduced to a minimum 40 Gy in 15 fractions over 3 weeks.)

    1. If the MGMT promoter in their tumor is known to be unmethylated, patients are not mandated to have received chemotherapy prior to participating in this trial
    2. If the MGMT promoter in their tumor is known to be methylated or the MGMT promoter methylation status is unknown at time of screening, patients must have received at least one chemotherapy regimen prior to participating in this trial
11. Patients with neoplastic lesions in the brainstem, cerebellum, or spinal cord; radiological evidence of active (growing) disease (active multifocal disease); extensive subependymal disease (tumor touching subependymal space is allowed); tumor crossing the midline or leptomeningeal disease
12. Patients on greater than 4 mg per day of dexamethasone within the 2 weeks prior to the 1st lerapolturev infusion via CED
13. Patients with worsening steroid myopathy (history of gradual progression of bilateral proximal muscle weakness, and atrophy of proximal muscle groups)
14. Patients with prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
15. Patients with active autoimmune disease requiring systemic immunomodulatory treatment within the past 3 months
16. Patients with known history of hypersensitivity to lomustine, dacarbazine, or any components of lomustine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients at each dose level who experienced a dose-limiting toxicity - Stage 1 | Up to 1 year
  Dose-limiting toxicities (DLTs) are defined as any of the following events that are possibly, probably, or definitely attributable to study treatment (i.e., lerapolturev) during dose escalation (Stage 1):
  * Any Grade 3 or any Grade 4 toxicity within 2 weeks, including cerebral edema or worsening neurologic symptoms
  * Any life-threatening event within 2 weeks
  * Treatment-related death at least possibly, probably, or definitely attributable to study treatment
  * Any grade 2 or higher serious cytokine release syndrome at least possibly, probably, or definitely attributable to study treatment, particularly those affecting vital organs (e.g., cardiac, hepatic, renal, CNS) occurring within 2 weeks of the infusion
Proportion of patients who experience an unacceptable toxicity - Stage 2 | Up to 1 year
  Unacceptable toxicity is defined as any of the following events that are possibly, probably, or definitely attributable to study treatment:
  * Any Grade 3 or any Grade 4 toxicity within 2 weeks, including cerebral edema or worsening neurologic symptoms
  * Any life-threatening event within 2 weeks
  * Treatment-related death at least possibly, probably, or definitely attributable to study treatment
  * Any grade 2 or higher serious cytokine release syndrome at least possibly, probably, or definitely attributable to study treatment, particularly those affecting vital organs (e.g., cardiac, hepatic, renal, CNS) occurring within 2 weeks of the infusion
Overall survival (OS) - Stage 2 | 2 years
  Median OS, where OS is defined as the time between randomization and death

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Median PFS, where PFS is defined as the time between randomization and initial failure (disease progression or death)

CONTACTS AND LOCATIONS:
Overall Officials: Madison Shoaf, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center — https://tischbraintumorcenter.duke.edu/
- See also: Duke Health — https://www.dukehealth.org/clinical-trials